CLINICAL TRIAL: NCT05026840
Title: Screening of GDM During COVID Pandemic in an Italian Setting. Comparison Between IADPSG and WHO '99 Criteria
Brief Title: GDM Screening During COVID Pandemic. IADPSG vs WHO '99 Criteria
Status: Completed | Type: Observational
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Rosario D'anna, full professor of obstetrics and gynecology, University of Messina
Other Study IDs: IADPSG vs WHO '99
Record Dates: First submitted 2021-08-27; First posted 2021-08-30 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: GDM Screening During COVID Pandemic; Comparison Between IADPSG vs WHO '99 Criteria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IADPSG
  Interventions: Procedure: GDM screening criteria
- WHO '99
  Interventions: Procedure: GDM screening criteria

INTERVENTIONS:
Procedure: GDM screening criteria — difference in risk factors and clinical outcomes between groups

SUMMARY:
All pregnant women who performed an OGTT following Italian Guidelines and then delivered at our University Hospital from march 2020 to march 2021 were prospectively enrolled in this study. Primary outcome of the study was the number of women to whom was diagnosed GDM with only the fasting glucose value (≥ 92 mg/dl), following Italian Diabetes Societies recommendations for COVID 19 pandemic period. In the same time, we prospectively collected the data of women who became diabetic following the criteria of WHO 1999 (fast glucose value ≥ 120 mg/dl, 2 hours later ≥ 140 mg/dl) still in use in some large countries like India. From the clinical charts, we reported the distribution of risk factors for GDM (maternal age ≥ 35 years, family history for diabetes type 2, ethnia, BMI ≥ 25, previous GDM) and clinical outcomes such as hypertensive disorders, preterm birth, macrosomia, intrauterine growth restriction and Caesarean section in emergency.

These data will be compared between the 2 groups consisting in those diagnosed with only IADPSG criteria versus those diagnosed with only WHO '99 criteria.

ELIGIBILITY:
Inclusion Criteria: Pregnant women who perform GDM screening -

Exclusion Criteria: Twin pregnancies

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All pregnant women who in a 12-month period perform GDM screening and then deliver at our University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
prevalence of women with a diagnosis of GDM following guidelines during COVID pamdemic | from march 2020 to march 2021
  evaluation of fast glucose level in the period recommended for GDM screening following Italian guidelines

SECONDARY OUTCOMES:
GDM diagnosis with IADPSG criteria versus WHO '99 criteria | from March 2020 to March 2021
  difference in risk factors and clinical outcomes between groups

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Messina, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] van-de-l'Isle Y, Steer PJ, Watt Coote I, Cauldwell M. Impact of changes to national UK Guidance on testing for gestational diabetes screening during a pandemic: a single-centre observational study. BJOG. 2021 Apr;128(5):917-920. doi: 10.1111/1471-0528.16482. Epub 2020 Oct 7. PMID 32888369
- [Derived] D'Anna R, Di Benedetto A, Palella S, Miceli A, Romeo P, Corrado F. Screening of GDM during COVID pandemic in an Italian setting: comparison between IADPSG and WHO '99 criteria. Diabetol Metab Syndr. 2022 Oct 31;14(1):164. doi: 10.1186/s13098-022-00936-4. PMID 36316733